CLINICAL TRIAL: NCT00872885
Title: A Randomized, Phase IIa Trial Evaluating the Safety and Efficacy of a New Centrally Acting Analgesic in Subjects With Moderate to Severe Pain Following Bunionectomy.
Brief Title: Bunionectomy Trial With GRT6005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 425965; KF5503/37 (Other: Sponsor)
Record Dates: First submitted 2009-03-24; First posted 2009-03-31 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Post Operative Pain
Keywords: analgesic; bunionectomy; surgery; post operative pain; single Hallux valgus repair
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): Dose 1
  Interventions: Drug: GRT6005
- B (Experimental): Dose 2
  Interventions: Drug: GRT6005
- C (Experimental): Dose 3
  Interventions: Drug: GRT6005
- D (Active Comparator): Morphine
  Interventions: Drug: Morphine
- E (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRT6005 — liquid formulation, 200 to 600 µg, single dose, one day
  Other Names: Morphine
  Arms: A; B; C
Drug: Morphine — 60 mg
  Arms: D
Drug: Placebo — single dosage
  Arms: E

SUMMARY:
The purpose of the trial is to determine whether the new centrally acting analgesic is effective in comparison to placebo and an active comparator (morphine).

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled to undergo primary unilateral first metatarsal bunionectomy

Exclusion Criteria:

* Contraindications to, or history of allergy or hypersensitivity to morphine, fentanyl, hydrocodone, acetaminophen, heparin, polyethylene glycol 400 USP-NF or any compound planned to be used during the anesthesia, or their excipients.
* Concomitant inflammatory disease.
* Life-long history of seizure disorder or epilepsy.
* Subjects with impaired renal function
* Subjects with impaired hepatic function
* Female subjects who are pregnant or breastfeeding.
* Resting pulse rate is <50bpm or >100 bpm after 5 minutes rest in supine position
* resting blood pressure after 5 minutes rest in supine position: Systolic blood pressure is <100mmHg or >140 mmHg Diastolic blood pressure is <60 mmHg or > 90 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity 2-10 hours after Investigational medicinal product intake. Pain assessments | 8 hours

SECONDARY OUTCOMES:
Amount of rescue medication | 24 hours
Adverse events | 24 hours
  Adverse Events reported by the participant as well as electrocardiogram, a measure of electrical activity of the heart and laboratory values
Time to first rescue medication | 24 hours
Patient Global Impression of Change | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: John Bothmer, Dr., Study Director — Grünenthal GmbH
Locations (1):
- Premier Research Group Ltd, Austin, Texas, United States